CLINICAL TRIAL: NCT03873636
Title: Altering Multitasking Behavior Using Low Current Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Nathan Ward, Assistant Professor, Tufts University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1611020
Record Dates: First submitted 2019-03-07; First posted 2019-03-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Change

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Stimulation (Experimental): Active stimulation of targeted brain regions involved in task-switching and dual-tasking.
  Interventions: Other: Stimulation via noninvasive brain stimulation systems
- Sham Stimulation (Sham Comparator): Sham stimulation of targeted brain regions involved in task-switching and dual-tasking.
  Interventions: Other: Stimulation via noninvasive brain stimulation systems

INTERVENTIONS:
Other: Stimulation via noninvasive brain stimulation systems — Active (at or below 2mA) stimulation targeting brain regions engaged in task-switching and dual-tasking for 30-40 minutes. Local IRB has determined the Soterix, Neuroelectrics, & Halo devices to be non-significant risk (NSR) devices via abbreviated investigational device exemption (IDE) procedure.

SUMMARY:
This study is designed to investigate multitasking deficits, with a particular interest in reducing costs related to dual-tasking (dividing attention between tasks) and task-switching (switching between tasks) using noninvasive brain stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to participate in non invasive brain stimulation research
* Must be a fluent English speaker
* Must be at least 18 years old
* Must be right-handed
* Must have normal or corrected-to-normal vision

Exclusion Criteria:

* Any history of complications with non invasive brain stimulation research
* Any metallic implants in head
* Any implanted internal or external electrical stimulation device
* Any adverse reaction to tDCS or other forms of low current brain stimulation
* Any history of seizure
* Any history of head injury
* Any illness that caused brain injury
* Any other brain-related condition
* Any diagnosis of neurological or psychiatric disorder
* A sensitive scalp

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-12-27 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Response accuracy | 4 hours
  Measuring accuracy (correct vs. incorrect answers) of responses to stimuli while dividing attention and switching between tasks
Response latency | 4 hours
  Measuring the amount of time (seconds) from when stimulus is presented to when participant answers prompt

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Ward, PhD, Principal Investigator — Tufts University
Locations (1):
- Tufts University, Medford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided